CLINICAL TRIAL: NCT02461628
Title: Innovative Partnership to Target Antimalarial Subsidies in the Retail Sector
Brief Title: Innovative Public-private Partnership to Target Subsidized Antimalarials in the Retail Sector (Aim 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Moi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00063384; 5R01AI110478 (NIH)
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Fever; Malaria
Keywords: Malaria; Antimalarial subsidy; Malaria rapid diagnostic test (RDT); Public-private partnership; Community health workers
MeSH Terms: conditions — Fever; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Malaria RDT & conditional voucher (Experimental): In the intervention arm, trained community health volunteers (CHVs) will offer eligible household members a free malaria rapid diagnostic test (RDT) and a voucher allowing the purchase of a qualified artemisinin combination therapy (ACT) at a reduced fixed price in the retail sector conditional on a positive test.
  Interventions: Behavioral: Malaria RDT & conditional voucher for ACT from retail sector
- Comparison Arm (No Intervention): Individuals in the comparison arm will only receive standard community health volunteer (CHV) visits.

INTERVENTIONS:
Behavioral: Malaria RDT & conditional voucher for ACT from retail sector — Trained community health volunteers will offer eligible household members free malaria rapid diagnostic tests and a voucher allowing the purchase of a qualified ACT at a reduced fixed price in the retail sector conditional on a positive test
  Arms: Malaria RDT & conditional voucher

SUMMARY:
The overall objective of this study is to evaluate the public health impact of targeted antimalarials subsidies through scale-up by determining the community-wide effects of targeting an antimalarial subsidy through a partnership between Community Health Volunteers (CHVs) and the private retail sector. The primary hypothesis to be tested is that offering a fixed-price voucher that reduces the cost for artemisinin combination therapy (ACT) purchase in the retail sector conditional on a positive malaria test (targeted subsidy) can improve uptake of testing for malaria and will increase the proportion of fevers tested for malaria before treatment. The study will be carried out in two sub-counties in Kenya with similar malaria burden but different access to health services; the investigators will use a cluster-randomized design to assign community units (CUs) in each sub-county to either an intervention or control arm. CHVs will be trained to use malaria rapid diagnostic tests (RDTs) to diagnose malaria in household members with documented or reported fever; households in intervention CUs will be informed of the intervention and encouraged to contact the CHV for any febrile illness in the home. There are minimal risks associated with receiving an RDT. Households with a positive RDT will be given a serialized voucher that will entitle the holder to purchase a quality assured ACT in the retail sector at a reduced, fixed price. The primary and secondary outcome measures will be compared at baseline and 12 months post-baseline through population-based surveying. The primary aim is to determine whether there is significant difference between the 2 study arms in the proportion of clients with fever who are tested prior to any treatment after adjusting for relevant covariates.

ELIGIBILITY:
INCLUSION CRITERIA

Intervention participation criteria:

* Client is older than 1 year
* Client has fever or history of fever or feeling unwell with a malaria-like illness within the last 2 days
* Client or their parent/legal guardian (if under 18) consents to participate

Cross sectional survey participation criteria:

* Household representative in the intervention or control arm
* At least one member in the respondent's household with a history of fever or feeling unwell with a malaria like illness within the last four weeks
* Respondent is older than 18 years

EXCLUSION CRITERIA

Intervention exclusion criteria:

* Client has signs of severe disease or other problem requiring immediate referral to a health facility
* Client has already visited a health facility, taken or purchased antimalarials for the current illness.

Cross sectional survey exclusion criteria:

• Households not in the intervention or control arms

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40340 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05-26 (Actual); Study Completion 2017-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy O'Meara, PhD, Principal Investigator — Duke University
Locations (1):
- Moi University, Eldoret, Kenya

REFERENCES:
- [Derived] Kirui J, Malinga J, Sang E, Ambani G, Abel L, Nalianya E, Namae J, Boyce M, Laktabai J, Menya D, O'Meara W. Supply-side and demand-side factors influencing uptake of malaria testing services in the community: lessons for scale-up from a post-hoc analysis of a cluster randomised, community-based trial in western Kenya. BMJ Open. 2023 Jun 26;13(6):e070482. doi: 10.1136/bmjopen-2022-070482. PMID 37369403
- [Derived] Prudhomme O'Meara W, Menya D, Laktabai J, Platt A, Saran I, Maffioli E, Kipkoech J, Mohanan M, Turner EL. Improving rational use of ACTs through diagnosis-dependent subsidies: Evidence from a cluster-randomized controlled trial in western Kenya. PLoS Med. 2018 Jul 17;15(7):e1002607. doi: 10.1371/journal.pmed.1002607. eCollection 2018 Jul. PMID 30016316
- [Derived] Laktabai J, Lesser A, Platt A, Maffioli E, Mohanan M, Menya D, Prudhomme O'Meara W, Turner EL. Innovative public-private partnership to target subsidised antimalarials: a study protocol for a cluster randomised controlled trial to evaluate a community intervention in Western Kenya. BMJ Open. 2017 Mar 20;7(3):e013972. doi: 10.1136/bmjopen-2016-013972. PMID 28320794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40340 participants signed consent. This is a cluster randomized trial with repeated measures; the repeated measures are independent cross-sectional samples of the population in each cluster. Participants at different time points are different participants who signed separate consent forms.
Pre-assignment Details: After enrollment, 7365 participants with a fever who received a malaria test from any source were approached to complete the survey. Only those 7365 participants are considered Started. Baseline data collection occurred before randomization of clusters to the arms.
Units Other Than Participants: Community Units
Groups:
- Malaria RDT & Conditional Voucher: In the intervention arm, trained community health volunteers (CHVs) will offer eligible household members a free malaria rapid diagnostic test (RDT) and a voucher allowing the purchase of a qualified ACT at a reduced fixed price in the retail sector conditional on a positive test.
  Malaria RDT & conditional voucher for ACT from retail sector: Trained community health volunteers will offer eligible household members free malaria rapid diagnostic tests and a voucher allowing the purchase of a qualified ACT at a reduced fixed price in the retail sector conditional on a positive test
Period: Overall Study
Arm/Group | Malaria RDT & Conditional Voucher | Comparison Arm
Started | 3733; 16 Community Units | 3632; 16 Community Units
Baseline Survey | 1038; 16 Community Units | 974; 16 Community Units
6 Month Survey | 814; 16 Community Units | 832; 16 Community Units
12 Month Survey | 882; 16 Community Units | 914; 16 Community Units
18 Month Survey | 995; 16 Community Units | 905; 16 Community Units
Completed | 3729; 16 Community Units | 3625; 16 Community Units
Not Completed | 4; 0 Community Units | 7; 0 Community Units
Not completed — Refused to complete survey | 4 | 7

BASELINE CHARACTERISTICS:
Population: All participants who completed the survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Malaria RDT & Conditional Voucher | Comparison Arm | Total
Number analyzed (Participants) | 3729 | 3625 | 7354
Age, Customized [Count of Participants; unit: Participants]
  Age: Under 5 years | 836 | 788 | 1624
  Age: 5 to 17 years | 1553 | 1480 | 3033
  Age: 18 years and above | 1340 | 1357 | 2697
  Age: Data missing | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2225 | 2198 | 4423
  Male | 1504 | 1427 | 2931
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 3729 | 3625 | 7354
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3729 | 3625 | 7354
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 3729 | 3625 | 7354

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Fever Who Receive a Malaria Test From Any Source
Time Frame: 6 months, 12 months, 18 months
Population: Subjects with fever who completed the survey at 6, 12, or 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Malaria RDT & Conditional Voucher | Comparison Arm
Number analyzed (Participants) | 2594 | 2573
Participants
  6 Months: number analyzed (Participants) | 783 | 810
  6 Months | 384 | 402
  12 Months: number analyzed (Participants) | 853 | 886
  12 Months | 443 | 391
  18 months: number analyzed (Participants) | 958 | 877
  18 months | 547 | 406

2. Secondary Outcome: Number of Participants Using ACT Who Had a Positive Test
Time Frame: 6 months, 12 months, 18 months
Population: Subjects who took AL and who completed the survey at 6, 12, or 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Malaria RDT & Conditional Voucher | Comparison Arm
Number analyzed (Participants) | 1865 | 1939
Participants
  6 Months: number analyzed (Participants) | 533 | 568
  6 Months | 234 | 305
  12 Months: number analyzed (Participants) | 596 | 679
  12 Months | 280 | 286
  18 months: number analyzed (Participants) | 736 | 692
  18 months | 426 | 302

3. Secondary Outcome: Number of Participants Using an ACT Who Did Not Have a Test
Time Frame: 6 months, 12 months, 18 months
Population: Subjects who took AL and who completed the survey at 6, 12, or 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Malaria RDT & Conditional Voucher | Comparison Arm
Number analyzed (Participants) | 1865 | 1939
Participants
  6 Months: number analyzed (Participants) | 533 | 568
  6 Months | 252 | 237
  12 Months: number analyzed (Participants) | 596 | 679
  12 Months | 260 | 363
  18 months: number analyzed (Participants) | 736 | 692
  18 months | 271 | 354

4. Secondary Outcome: Number of Subjects Who Received a Correct Dose of AL (Artemether Lumefantrine)
Description: Denominator is all those who took AL. Artemether lumefantrine is one type of ACT.
Time Frame: 6 months, 12 months, 18 months
Population: Subjects who received AL and completed the survey at 6, 12, or 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Malaria RDT & Conditional Voucher | Comparison Arm
Number analyzed (Participants) | 1783 | 1832
Participants
  6 Months: number analyzed (Participants) | 515 | 547
  6 Months | 338 | 352
  12 Months: number analyzed (Participants) | 550 | 614
  12 Months | 376 | 391
  18 months: number analyzed (Participants) | 718 | 671
  18 months | 496 | 410

5. Secondary Outcome: Number of Subjects With Fever That Received Correct Treatment
Description: The number of people with fever that report receiving correct treatment with regards to malaria (i.e., received an RDT test and took ACTs if the result was positive, or did not take ACTs if the test result was negative).
Time Frame: 6 months, 12 months, 18 months
Population: Subjects with fever who completed the survey at 6, 12, or 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Malaria RDT & Conditional Voucher | Comparison Arm
Number analyzed (Participants) | 2594 | 2573
Participants
  6 Months: number analyzed (Participants) | 783 | 810
  6 Months | 309 | 340
  12 Months: number analyzed (Participants) | 853 | 886
  12 Months | 344 | 306
  18 months: number analyzed (Participants) | 958 | 877
  18 months | 462 | 321

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse event data were collected on subjects who completed the survey at baseline, 6, 12, or 18 months.
Arm/Group | Malaria RDT & Conditional Voucher | Comparison Arm
All-Cause Mortality (participants affected / at risk) | 0/3729 | 0/3625
Serious Adverse Events (participants affected / at risk) | 0/3729 | 0/3625
Other Adverse Events (participants affected / at risk) | 0/3729 | 0/3625

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT02461628/Prot_SAP_000.pdf